CLINICAL TRIAL: NCT02564887
Title: Pilot Study to Improve Therapeutic Outcomes for Dysphagia After Radiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment goals not met in efficient timeframe.
Sponsor: Jonas Johnson (Other)
Responsible Party: Sponsor-Investigator, Jonas Johnson, Professor and Chairman, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRO15080566
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Dysphagia; Oral Pharyngeal Cancer
Keywords: dysphagia; oral pharyngeal cancer; Iowa Oral Performance Instrument (IOPI); IOPI
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Therapy Only (Other): Standard of care therapy for qualifying population (with opportunity to "crossover" and be assigned to the IOPI device if so desired after initial 8 week standard of care therapy completion.
  Interventions: Device: Iowa Oral Performance Instrument
- Traditional Therapy with IOPI (Experimental): Standard of care therapy plus the addition of the IOPI instrument
  Interventions: Device: Iowa Oral Performance Instrument

INTERVENTIONS:
Device: Iowa Oral Performance Instrument — the IOPI device is being used to increase tongue strength and endurance
  Other Names: IOPI

SUMMARY:
Patients with head and neck cancer treated with chemoradiation, often develop a treatment associated dysphagia. The common complaint is foods sticking in the pharynx. This study seeks to test the Iowa Oral Performance Instrument (IOPI) in the management of treatment induced dysphagia following chemoradiation for oral, pharyngeal, laryngeal, hypopharyngeal cancer. This pilot study seeks to compare standard exercise therapy plus IOPI to standard exercise alone to determine if recovery is enhanced and to determine if rate of recovery is accelerated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with oral, oropharyngeal, hypopharyngeal or laryngeal cancer having non-surgical treatment with chemoradiation, or radiation therapy alone, resulting in treatment associated dysphagia.

Exclusion Criteria:

* unable to adhere to assigned therapy program due to cognitive deficits
* surgical treatment for head and neck cancer
* unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-01; Primary Completion 2019-01-31 (Actual); Study Completion 2019-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Traditional Therapy Only | Traditional Therapy With IOPI
Started | 16 | 10
Completed | 10 | 10
Not Completed | 6 | 0
Not completed — Lost to Follow-up | 6 | 0

BASELINE CHARACTERISTICS:
Population: Information is reported for the 20 participants who have completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Therapy Only | Traditional Therapy With IOPI | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Full Range); unit: years] | 62.7 [52 to 77] | 62 [36 to 81] | 62 [36 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 26
Tongue Strength (kPa) [Mean (Full Range); unit: kPa] | 44.5 [27 to 63] | 41.4 [13 to 73] | 42.95 [13 to 73]

OUTCOME MEASURES:

1. Primary Outcome: Tongue Pressure Generation (i.e. Tongue Strength) in Kilopascals (kPa) Using the IOPI Device
Description: Change in tongue strength from baseline measurements; 2nd measurement collected post treatment (approximately 8 weeks from baseline)
Time Frame: 8 weeks
Measure: Mean (Full Range); unit: kPa
Groups:
- Traditional Therapy Only: Standard of care therapy for qualifying population (with opportunity to "crossover" and be assigned to the IOPI device if so desired after initial 8 week standard of care therapy completion.
  Iowa Oral Performance Instrument: the IOPI device is being used to increase tongue strength and endurance
  Tongue strength was measured pre- and post-treatment with the Iowa Oral performance Instrument which measures linguapalatal pressure/force generation in kilopascals of pressure.
- Traditional Therapy With IOPI: Standard of care therapy plus the addition of the IOPI instrument
  Iowa Oral Performance Instrument: the IOPI device is being used to increase tongue strength and endurance
  Tongue strength was measured pre- and post-treatment with the Iowa Oral performance Instrument which measures linguapalatal pressure/force generation in kilopascals of pressure.
Arm/Group | Traditional Therapy Only | Traditional Therapy With IOPI
Number analyzed (Participants) | 10 | 10
kPa | 7.9 [0 to 13] | 5.1 [-4 to 23]

2. Secondary Outcome: Airway Protection During Swallowing
Description: Penetration-aspiration scale score of the modified barium swallow (MBS) data for small, thin liquids Scores are determined primarily by the depth to which material passes in the airway and by whether or not material entering the airway is expelled.
  Minimum 1 Maximum 8 Lower is better The score being evaluated is an absolute score at the time of collection and not the change over time.
Time Frame: 8 week
Population: Not all participants were evaluated using a modified barium swallow test. Reasons that a participant did not perform the MBS, would be safety (the clinician did not feel that is was safe for the participant to undergo the MBS) or not indicated (an MBS was not clinically indicated at that time). Only completed MBS tests were evaluated.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Traditional Therapy Only | Traditional Therapy With IOPI
Number analyzed (Participants) | 4 | 9
score on a scale | 4.875 [2 to 6.5] | 4.56 [1 to 8]

3. Secondary Outcome: Change Over Time of Pharyngeal Residue After Swallowing
Description: The change in pharyngeal retention measured using the normalized residue ratio scale (NRR) is being assessed.
  The NRR quantifies the amount of residue remaining in the valleculae and pyriform sinuses after a swallow as a ratio of the total area of each of these two pharyngeal spaces.
  Value represents the area of space that is occupied by barium at the end of a swallow.
  The change from baseline to 8 weeks is documented.
  A positive change (+) is worsening of symptoms. A negative change (-) is bettering of symptoms.
Time Frame: 8 week
Population: While the Traditional Therapy Only and the Traditional Therapy with IOPI groups each contain n=10 participants, only 6 swallowing evaluations underwent evaluation for this particular measure.
  Detailed swallowing evaluations were only performed in participants who were felt to be "safe" to undergo the evaluations.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Traditional Therapy Only | Traditional Therapy With IOPI
Number analyzed (Participants) | 6 | 6
units on a scale
  Pyriform | .0160 [-.0013 to .0587] | .0105 [-.0001 to .0310]
  Vallecula | -.0268 [-.0431 to .0131] | -.0589 [-.2007 to .03]

4. Secondary Outcome: Swallowing Impairment-Self Report
Description: Patient perceived outcome measure related to their view of their swallowing problem/difficulties at that point in time.
  Eating Assessment Tool (EAT-10). Minimum score 0 Maximum score 40 Higher score is worse Number reported is final overall score
Time Frame: 8 week
Measure: Mean (Full Range); unit: score on scale
Arm/Group | Traditional Therapy Only | Traditional Therapy With IOPI
Number analyzed (Participants) | 10 | 10
score on scale | 14.4 [3 to 24] | 15.5 [3 to 34]

5. Secondary Outcome: Swallowing Impairment
Description: visual analog scale related to patient perceived swallowing impairment at that point in time.
  Minimum - 0 Maximum - 100 Higher is worse Score reported is the overall score at that time and not a change from baseline.
Time Frame: 8 week
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Traditional Therapy Only | Traditional Therapy With IOPI
Number analyzed (Participants) | 10 | 10
score on a scale | 31.1 [5 to 60] | 30.5 [0 to 80]

6. Secondary Outcome: Swallowing Impairment-Objective
Description: functional oral intake scale (FOIS) The Functional Oral Intake Scale is an ordinal scale that is used to assess the current status and meaningful change in the oral intake.
  Minimum - 1 Maximum - 7 Higher is better Score reported is the overall score at that point in time and not a change from baseline.
Time Frame: 8 week
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Traditional Therapy Only | Traditional Therapy With IOPI
Number analyzed (Participants) | 10 | 10
score on a scale | 5.5 [2 to 7] | 5.2 [2 to 7]

ADVERSE EVENTS:
Time Frame: 2 years, 8 months
Description: No adverse events, as defined by the University of Pittsburgh Institutional Review Board, occurred during the course of this research.
Arm/Group | Traditional Therapy Only | Traditional Therapy With IOPI
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/10
Other Adverse Events (participants affected / at risk) | 0/16 | 0/10

LIMITATIONS AND CAVEATS:
Enrollment for the study was lower than anticipated. This may be attributed to decreased availability of dedicated research personnel trained in the use of the IOPI device. Greater resources are now available for future studies in this area.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT02564887/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT02564887/Prot_SAP_001.pdf